CLINICAL TRIAL: NCT00711256
Title: Sunscreen Removal by Clothing Meassured in Vivo. Sun Protection Factor Persistence During a Day Indoor Without Physical Activity. Does Sunscreen Reduce Vitamin D?
Brief Title: Sunscreen: Persistence of Sun Protection Factor and the Influence on Vitamin D
Acronym: sunscreen
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Bispebjerg Hospital. Dr. Hans Christian Wulf, Bispebjerg Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: H-B-2007-120
Record Dates: First submitted 2008-07-07; First posted 2008-07-08 (Estimated); Last update posted 2008-07-08 (Estimated); Status verified 2008-04

CONDITIONS: Vitamin D Production in the Skin; Sunscreen Persistence
Keywords: Sunscreen; Application; Vitamin D; Sun protection factor; Clothing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): No sunscreen applied
  Interventions: Radiation: UVB light
- 2 (Active Comparator): Sunscreen applied 0.5 mg/cm2
  Interventions: Radiation: UVB light
- 3 (Active Comparator): Sunscreen applied 1mg/cm2
  Interventions: Radiation: UVB light
- 4 (Active Comparator): Sunscreen applied 2mg/cm2
  Interventions: Other: sunscreen MATAS sunlotion SPF 8; Radiation: UVB light

INTERVENTIONS:
Other: sunscreen MATAS sunlotion SPF 8
  Other Names: MATAS sollotion. Matas Denmark, 3400 Alleroed
  Arms: 4
Radiation: UVB light — duration 4 times 1 minute radiation on the trunk.

SUMMARY:
The investigators want to investigate whether sunscreen is removed by clothing and to what extend when the amount of sunscreen applied varies.Does clothing reduce the SPF when clothes are put on 20, 8, or 4 minutes after sunscreen application? The investigators also want to investigate the persistence of sunscreen during eight hours indoor. How much does the SPF reduces? Furthermore, we want to investigate whether sunscreen in the layers 2, 1, and 0.5 mg/cm2 reduce the vitamin D production in the skin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participants.
* > 18 years.
* Skin type I, II, and III.

Exclusion Criteria:

* Pregnancy.
* Medicin use.
* Skin or other diseases.
* The participants must not have been in solarium or gotten sun on their trunks in the 3 months before the study start and during the study.
* Skin types IV and above.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-07; Primary Completion 2008-08 (Estimated); Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
vitamin D (nmol) meassured in a blood sample. | 5 days after sunscreen use and UV light exposure

CONTACTS AND LOCATIONS:
Locations (1):
- Bispebjerg Hospital, Copenhagen, KBH NV, Denmark

REFERENCES:
- [Derived] Beyer DM, Faurschou A, Philipsen PA, Haedersdal M, Wulf HC. Sun protection factor persistence on human skin during a day without physical activity or ultraviolet exposure. Photodermatol Photoimmunol Photomed. 2010 Feb;26(1):22-7. doi: 10.1111/j.1600-0781.2009.00479.x. PMID 20070835